CLINICAL TRIAL: NCT00430963
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Multicenter Trial With an Open-label Extension Period to Investigate the Efficacy and Safety of IncobotulinumtoxinA (Xeomin), Free of Complexing Proteins, in the Treatment of Glabellar Frown Lines
Brief Title: IncobotulinumtoxinA (Xeomin) Versus Placebo in the Treatment of Glabellar Frown Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 60201-0520/1
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo to IncobotulinumtoxinA (Xeomin) powder for solution for injection; dose: one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl, corresponding to total placebo volume 0.5 mL; mode of administration: intramuscular injection
  Interventions: Drug: Placebo
- IncobotulinumtoxinA (Xeomin) (20 Units) (Experimental): IncobotulinumtoxinA (Xeomin), also known as 'NT 201' or 'Botulinum toxin type A (150 kD), free from complexing proteins' (active ingredient: Clostridium Botulinum neurotoxin type A free from complexing proteins) powder for solution for injection; dose: one injection session of solution, prepared by reconstitution of powder with 0.9% sodium chloride (NaCl), 20 units, total volume 0.5 mL, mode of administration: intramuscular injection
  Interventions: Drug: IncobotulinumtoxinA (Xeomin) (20 Units)

INTERVENTIONS:
Drug: IncobotulinumtoxinA (Xeomin) (20 Units)
  Arms: IncobotulinumtoxinA (Xeomin) (20 Units)
Drug: Placebo
  Arms: Placebo

SUMMARY:
IncobotulinumtoxinA (Xeomin) is a botulinum toxin type A preparation free of complexing proteins, i.e. free of proteins other than the active toxin. Injected into the muscle, IncobotulinumtoxinA (Xeomin) causes local weakening. Botulinum toxin type A is widely used for aesthetic treatment of facial lines. This study investigated the efficacy and safety of IncobotulinumtoxinA (Xeomin) in the treatment of glabellar frown lines compared to placebo. The study consisted of a Main Period and an Open-Label Extension [OLEX] Period of 120 days each.

ELIGIBILITY:
Inclusion Criteria:

•Moderate to severe glabellar frown lines

Exclusion Criteria:

* Previous insertion of permanent material in the glabellar area
* Neuromuscular function disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Investigator's assessment according to the Facial Wrinkle Scale (FWS) | Day 30
  Responder: FWS score of 0 or 1.
Patient's global assessment | Day 30
  Responder: subjects with a score of at least 2+.

SECONDARY OUTCOMES:
Investigator's assessment according to FWS | Day 7, 60, 90, and 120
  Responder: FWS score of 0 or 1.
Patient's global assessment | Day 7, 60, 90, and 120
  Responder: subjects with a score of at least 2+.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (1):
- Merz Pharmaceuticals GmbH, Frankfurt, Germany